CLINICAL TRIAL: NCT02216903
Title: Respiratory Motion Related Ablation Gap and Clinical Outcome After Catheter Ablation for Atrial Fibrillation
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2014-0502
Record Dates: First submitted 2014-08-13; First posted 2014-08-15 (Estimated); Last update posted 2019-03-27 (Actual); Status verified 2018-02

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation, sleep apnea
MeSH Terms: conditions — Atrial Fibrillation; Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Yonsei AF Cohort: Patients with atrial fibrillation who undergoing catheter ablation of atrial fibrillation

SUMMARY:
This is the evaluation which is associated with apnea symptom, one of the recurrence factors, after AF ablation to patients who diagnosed AF.

This is the evaluation which is associated with excessive respiration exercise during AF ablation to patients who diagnosed AF.

This is the evaluation which is associated with excessive respiration exercise to make a gap during AF ablation to patients who diagnosed AF.

ELIGIBILITY:
Inclusion Criteria:

1. age 20~80
2. Left atrium size <55mm

Exclusion Criteria:

1. Permeant AF which is uncontrolled by cardioverting
2. Valvular AF (mitral stenosis> grade 2, mitral valvuloplasty)
3. Structural heart disease which is necessary operation to be healed.
4. The patients who had history of ablation or maze operation
5. The patients who have abnormal respiration by spinal or chest modification.
6. accompany Severe disease in present
7. Under age <20

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with atrial fibrillation who undergoing catheter ablation in Yonsei Cardiovascular hospital, Yonsei university health system, Seoul, Korea.
Sampling Method: Non-Probability Sample
Enrollment: 510 (Actual)
Dates: Start 2014-08; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Clinical recurrence of atrial fibrillation (AF) after catheter ablation | after 90 days of catheter ablation and thereafter
  We defined recurrence of AF as any episode of AF or atrial tachycardia lasting longer than 30 sec. Any ECG documentation of AF recurrence after 3 months was diagnosed as clinical recurrence.

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea